Soft Tissue Augmentation by Xenogeneic Collagen Matrix Versus Subepithelial Connective Tissue Grant Co

# Statistical Analysis Plan

Document Type: Statistical Analysis Plan

NCT Number: (To be assigned) Document Date: July 3, 2021

Submitted by: Mohamed Omar Ismail PhD Candidate Faculty of Dentistry Minia University

## 1. Study Identification

- Protocol ID: 505/2021
- Sponsor: Minia University
- Investigator: Mohamed Omar Ismail, PhD Candidate

#### 2. Study Objectives

- To compare the clinical outcomes of xenogeneic collagen matrix (XCM) and subepithelial connective

### 3. Endpoints

- Primary Endpoint: Change in peri-implant soft tissue thickness at 12 months (in mm).

## 4. Study Design Summary

- Randomized controlled trial with two parallel arms.
- 20 patients (10 per group), assigned to either SCTG or XCM group.
- Outcome assessed by a blinded evaluator.

## 5. Sample Size Justification

- Based on clinical experience and prior literature, a sample size of 10 per group was determined to

#### 6. Statistical Methods

- Descriptive statistics (mean, SD) will be used for baseline characteristics.
- Independent Samples T-test will be used to compare changes in soft tissue thickness between gro
- Significance level set at p < 0.05.
- Confidence interval: 95%

### 7. Missing Data Handling

- Missing values will be managed using pairwise deletion. No imputation methods are planned.

#### 8. Software to be Used

- Statistical analysis will be conducted using SPSS version 25 (IBM Corp.).

#### 9. Data Presentation

- Data will be presented in tables (means ± SD).
- Results will be illustrated using bar charts to compare primary outcomes.